CLINICAL TRIAL: NCT06150391
Title: Randomized Controlled Trial of a Dichoptic Gabor Videogame Program to Improve Visual Function in Children With Amblyopia
Brief Title: Evaluation of Amblyopia Protocols Using a Dichoptic Gabor Videogame Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Merida (Other)
Collaborators: VisionaryTool, S.L. (Unknown)
Responsible Party: Principal Investigator, Maria Perez-Benito, Dr., Hospital de Merida
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEI 046/23
Record Dates: First submitted 2023-11-13; First posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Amblyopia
Keywords: amblyopia; perceptual learning; dichoptic therapy; visual acuity
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Intervention Model Description: Participants will be divided in two groups: GA, 60 participants without previous occlusion treatment; GB, 60 participants with previous occlusion or penalization.
  In GA, participants will be assigned to an Experimental subgroup (GA-E) or to a Control subgroup (GA-C). GA-E volunteers will be prescribed computer-based exercises (Visionary). GA-C patients will be prescribed occlusion.
  In GB, all participants will receive occlusion. There will be two subgroups, Experimental (GB-E) and Control (GB-C), and both will be prescribed exercises using Visionary. In GB-E the computer will adjust Gabor patches frequency to visual acuity, as normal; but in GB-C Gabor frequencies will always be low.
  Importantly, those patients with deviations (10 to 25 prismatic diopters) will be assigned to experimental or treatment subgroups following an independent randomization.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Ophthalmologists at the Pediatric Ophthalmologic Unit (Care Provider and Outcomes Assessor) will decide if volunteers meet inclusion criteria. They will assign the patient to GA or GB. They will be responsible for final and after treatment visual evaluations.
  The Quality Service of the Merida Hospital (Investigator) will randomize GA and GB volunteers into treatment or control subgroups. This service will be responsible for the custody of documentation and the statistical final analysis.
  Visionary team (Investigator) will communicate the patient about the treatment (occlusion or Visionary software, or both).
  Optometrists at the Pediatric Ophthalmologic Unit (Outcomes Assessor) will oversee BCVA and stereoacuity measurements during treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group GA-E. Patients without previous occlusion o penalization treatment - Experimental (Experimental): GA-E volunteers (experimental) will be prescribed home therapy using computer-based exercises (Visionary) for 12 weeks, five days week, ½ half hour per day. Visionary target frequencies will be adjusted, considering BCVA, each three weeks. Contrast of Gabor patch frequencies will be adjusted to match patient contrast sensitivity thresholds.
  In case BCVA does not improve at least 2 lines in two consecutive visits (6 weeks), patients will change to GA-C.
  Interventions: Device: Visionary: computer exercises using dichoptic Gabor Patches and band-filtered noise masks
- Group GA-C. Patients without previous occlusion o penalization treatment - Control (Active Comparator): GA-C patients (control) will be prescribed occlusion following Pediatric Eye Disease Investigation Group (PEDIG) criteria: 2 hours for mild and moderate amblyopia or 6 hours for severe amblyopia. Patients will receive a calendar to track patching accomplishment.
  In case BCVA does not improve at least 2 lines in two consecutive visits (6 weeks), patients will change to GA-E.
  Interventions: Device: Patching
- Group GB-E. Patients with previous occlusion o penalization treatment - Experimental (Experimental): GB-E volunteers will receive occlusion following PEDIG criteria and will be prescribed home therapy using Visionary. Patients will receive a calendar to track patching accomplishment.
  Visionary target frequencies will be adjusted, considering BCVA, each three weeks.
  Interventions: Device: Visionary: computer exercises using dichoptic Gabor Patches and band-filtered noise masks; Device: Patching
- Group GB-C. Patients with previous occlusion o penalization treatment - Control (Active Comparator): GB-C volunteers will receive occlusion following PEDIG criteria and will be prescribed home therapy using Visionary. Patients will receive a calendar to track patching accomplishment.
  Visionary target frequencies will always be low, no matter patient VA.
  In case BCVA does not improve at least 2 lines in two consecutive visits (6 weeks), patients will be move to GB-E.
  Interventions: Device: Visionary: computer exercises using dichoptic Gabor Patches and band-filtered noise masks; Device: Patching

INTERVENTIONS:
Device: Visionary: computer exercises using dichoptic Gabor Patches and band-filtered noise masks — Visionary exercises are computer gammified activities that run on a computer with internet connection to facilitate home therapy. Patient must wear anaglyph glasses. Visual stimuli consists in dichoptic Gabor Patches presented to the amblyopic eye. Frequency is adjusted to actual patient visual acuity, and contrast to actual patient performance (contrast sensitivity). A band-filtered noise mask at the same frequency than the Gabor patch is presented to the fellow eye in certain ocassions.
  Arms: Group GA-E. Patients without previous occlusion o penalization treatment - Experimental; Group GB-C. Patients with previous occlusion o penalization treatment - Control; Group GB-E. Patients with previous occlusion o penalization treatment - Experimental
Device: Patching — PEDIG (Pediatric Eye Disease Investigator Group) recommended amblyopia treatment. Consist on covering a child's better-seeing eye with a patch for 2 hours per day for mild and moderate amblyopia or 6 hours per day for severe amblyopia
  Arms: Group GA-C. Patients without previous occlusion o penalization treatment - Control; Group GB-C. Patients with previous occlusion o penalization treatment - Control; Group GB-E. Patients with previous occlusion o penalization treatment - Experimental

SUMMARY:
Interest in developing alternative methods for the treatment of amblyopia (lazy eye) has long been a topic of interest among clinicians and researchers. Occlusion or penalization of fellow eye do not always provide the desired visual acuity improvement. Moreover, occlusion is associated with a high risk of recurrence and non-compliance. Here, it is presented a protocol of a randomized clinical trial to evaluate the safety and clinical efficacy of a novel home-based system, based on a computer game.

The goal of this prospective clinical trial is to compare in visual acuity improvements in patients with amblyopia, following conventional patching therapy or this novel computer-based therapy.

The main questions it aims to answer are:

* Does computer-based therapy equal or improve patching therapy? Can it be used as an alternative to patching?
* Does computer-based therapy used in combination with pathching solve amblyopia when patching fails alone (persistent amblyopia)?

Participants will be divided in two groups according to the previous occlusion o penalization of fellow eye. Both groups will be divided in two subgroups, experimental and control. Researchers will compare subgroups outcomes in order to asses this novel approach.

DETAILED DESCRIPTION:
Amblyopia is a common neurodevelopmental abnormality that results in physiological alterations of the visual pathways and impaired vision in one eye or, less commonly, in both.Disruption of normal visual development early in life may result in perceptual, oculomotor and clinical abnormalities such as instability of fixation, anomalous retinal correspondence, and lack of stereoacuity.Amblyopia has a prevalence of around 2-4% in children and is associated with refractive error (anisometropia or isometropia) and strabismus.

The Pediatric Eye Disease Investigator Group (PEDIG) has produced several studies that analyze the most effective therapies for amblyopic eye. The gold standard treatment prescribed for this condition combines spectacle correction of the refractive error with penalization and/or occlusion of the dominant eye

Interest in developing alternative methods for the treatment of amblyopia (lazy eye) has long been a topic of interest among clinicians and researchers. Occlusion or penalization of fellow eye do not always provide the desired visual acuity improvement. Moreover, occlusion is associated with a high risk of recurrence and non-compliance.

This randomized clinical trial is designed to evaluate the safety and clinical efficacy of a novel home-based system, based on a computer activity that uses dichoptic Gabor Patches and band-filtered noise masks. It combines the concepts of perceptual learning, dichoptic training, home based therapy and gamification.

The goal of this prospective clinical trial is to compare in visual acuity improvements in patients with amblyopia, following conventional patching therapy or this novel computer-based therapy.

The main questions it aims to answer are:

* Does computer-based therapy equal or improve patching therapy? Can it be used as an alternative to patching?
* Does computer-based therapy used as coadjuvant to pathching solve amblyopia in patients where patching fails alone (persistent amblyopia)?

Participants will be divided in two groups according to the previous occlusion o penalization of fellow eye. Both groups will be divided in two subgroups, experimental and control. Researchers will compare subgroups outcomes in order to asses if this novel approach may lead to greater improvements in vision performance in amblyopic children as substitution of occlusion treatment in novel amblyopia or as coadjutant in persistent amblyopia.

ELIGIBILITY:
Inclusion Criteria:

* The sample will be made up of children with amblyopia from 4 to 12 years old (amblyopia will be defined as the best corrected visual acuity less o equal to 0.8 in decimal units or > 2 lines of difference between both eyes). Strabismus inclusion criteria will be < 25 prismatic diopters, with a deviation ≥ 2 prismatic diopters.

Exclusion Criteria:

* Subjects with nystagmus, ocular pathology o cognitive delay will be excluded.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
BCVA Best Corrected Visual Acuity | Treatment will last 12 weeks, with BCVA measurements every 2 weeks. The stability control post treatment will last 12 months, with BCVA controls at 3, 6 and 12 months.
  Best Corrected Visual Acuity is the measurement of the ability to distinguish shapes and the details of objects at a given distance wearing full refraction. Different optotipes are used to measure clinically this ability (e.g. Snellen E, ETDRS, etc.). Refraction must be calculated under cyclopegia following PEDIG criteria. Crowding bars can be added to the optotypes.
  In this study, amblyopic eye BCVA will be measured using visual acuity chart ETDRS whitout crowding bars, in logarithmic scale.

SECONDARY OUTCOMES:
Stereoacuity | Treatment will last 12 weeks, with stereoacuity measurements every 2 weeks. The stability control post treatment will last 12 months, with stereoacuity controls at 3, 6 and 12 months.
  In this stuty Randot Preschool Stereoacuity Test (Stereo Optical, Inc., Chicago, USA) will be used to asses stereoacuity in arc seconds. This is a random dot stereogram that measures global stereopsis (or cyclopean stereopsis) and does not contain monocular cues. Stereoacuity is measured at a constant distance of 40 cm.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Calderon-Gonzalez, Lic, Study Chair — VisionaryTool, S.L.; Juan A. Portela-Camino, PhD, Study Chair — VisionaryTool, S.L.; Santiago Martin-Gonzalez, PhD, Study Chair — VisionaryTool, S.L.; Maria Perez-Benito, Dra, Principal Investigator — Hospital de Merida; Esther Alvarez-Martin, Dra, Study Chair — Hospital de Merida
Locations (1):
- Servicio de Oftalmología del Hospital de Merida, Mérida, Extremadura, Spain

REFERENCES:
- [Background] Verghese P, McKee SP, Levi DM. Attention deficits in Amblyopia. Curr Opin Psychol. 2019 Oct;29:199-204. doi: 10.1016/j.copsyc.2019.03.011. Epub 2019 Mar 22. PMID 31030000
- [Background] Fu Z, Hong H, Su Z, Lou B, Pan CW, Liu H. Global prevalence of amblyopia and disease burden projections through 2040: a systematic review and meta-analysis. Br J Ophthalmol. 2020 Aug;104(8):1164-1170. doi: 10.1136/bjophthalmol-2019-314759. Epub 2019 Nov 8. PMID 31704700
- [Background] Chen AM, Cotter SA. The Amblyopia Treatment Studies: Implications for Clinical Practice. Adv Ophthalmol Optom. 2016 Aug;1(1):287-305. doi: 10.1016/j.yaoo.2016.03.007. No abstract available. PMID 28435934
- [Background] Birch EE. Amblyopia and binocular vision. Prog Retin Eye Res. 2013 Mar;33:67-84. doi: 10.1016/j.preteyeres.2012.11.001. Epub 2012 Nov 29. PMID 23201436
- [Background] Buckle M, Billington C, Shah P, Ferris JD. Treatment outcomes for amblyopia using PEDIG amblyopia protocols: a retrospective study of 877 cases. J AAPOS. 2019 Apr;23(2):98.e1-98.e4. doi: 10.1016/j.jaapos.2018.12.007. Epub 2019 Mar 30. PMID 30935990
- [Background] GIBSON EJ. Perceptual learning. Annu Rev Psychol. 1963;14:29-56. doi: 10.1146/annurev.ps.14.020163.000333. No abstract available. PMID 13947716
- [Background] Rodan A, Candela Marroquin E, Jara Garcia LC. An updated review about perceptual learning as a treatment for amblyopia. J Optom. 2022 Jan-Mar;15(1):3-34. doi: 10.1016/j.optom.2020.08.002. Epub 2020 Nov 24. PMID 33243673
- [Background] Polat U, Ma-Naim T, Belkin M, Sagi D. Improving vision in adult amblyopia by perceptual learning. Proc Natl Acad Sci U S A. 2004 Apr 27;101(17):6692-7. doi: 10.1073/pnas.0401200101. Epub 2004 Apr 19. PMID 15096608
- [Background] Polat U, Ma-Naim T, Spierer A. Treatment of children with amblyopia by perceptual learning. Vision Res. 2009 Oct;49(21):2599-603. doi: 10.1016/j.visres.2009.07.008. Epub 2009 Jul 19. PMID 19622368
- [Background] Barollo M, Contemori G, Battaglini L, Pavan A, Casco C. Perceptual learning improves contrast sensitivity, visual acuity, and foveal crowding in amblyopia. Restor Neurol Neurosci. 2017;35(5):483-496. doi: 10.3233/RNN-170731. PMID 28800339
- [Background] Levi DM, Li RW. Perceptual learning as a potential treatment for amblyopia: a mini-review. Vision Res. 2009 Oct;49(21):2535-49. doi: 10.1016/j.visres.2009.02.010. Epub 2009 Feb 27. PMID 19250947
- [Background] Chen PL, Chen JT, Fu JJ, Chien KH, Lu DW. A pilot study of anisometropic amblyopia improved in adults and children by perceptual learning: an alternative treatment to patching. Ophthalmic Physiol Opt. 2008 Sep;28(5):422-8. doi: 10.1111/j.1475-1313.2008.00588.x. PMID 18761479
- [Background] Stewart CE, Moseley MJ, Stephens DA, Fielder AR. Treatment dose-response in amblyopia therapy: the Monitored Occlusion Treatment of Amblyopia Study (MOTAS). Invest Ophthalmol Vis Sci. 2004 Sep;45(9):3048-54. doi: 10.1167/iovs.04-0250. PMID 15326120
- [Background] Baker DH, Meese TS, Mansouri B, Hess RF. Binocular summation of contrast remains intact in strabismic amblyopia. Invest Ophthalmol Vis Sci. 2007 Nov;48(11):5332-8. doi: 10.1167/iovs.07-0194. PMID 17962490
- [Background] Li SL, Jost RM, Morale SE, Stager DR, Dao L, Stager D, Birch EE. A binocular iPad treatment for amblyopic children. Eye (Lond). 2014 Oct;28(10):1246-53. doi: 10.1038/eye.2014.165. Epub 2014 Jul 25. PMID 25060850
- [Background] Birch EE, Li SL, Jost RM, Morale SE, De La Cruz A, Stager D Jr, Dao L, Stager DR Sr. Binocular iPad treatment for amblyopia in preschool children. J AAPOS. 2015 Feb;19(1):6-11. doi: 10.1016/j.jaapos.2014.09.009. PMID 25727578
- [Background] Manh VM, Holmes JM, Lazar EL, Kraker RT, Wallace DK, Kulp MT, Galvin JA, Shah BK, Davis PL; Pediatric Eye Disease Investigator Group. A Randomized Trial of a Binocular iPad Game Versus Part-Time Patching in Children Aged 13 to 16 Years With Amblyopia. Am J Ophthalmol. 2018 Feb;186:104-115. doi: 10.1016/j.ajo.2017.11.017. Epub 2017 Nov 28. PMID 29196184
- [Background] Kelly KR, Jost RM, Dao L, Beauchamp CL, Leffler JN, Birch EE. Binocular iPad Game vs Patching for Treatment of Amblyopia in Children: A Randomized Clinical Trial. JAMA Ophthalmol. 2016 Dec 1;134(12):1402-1408. doi: 10.1001/jamaophthalmol.2016.4224. PMID 27832248
- [Background] Pediatric Eye Disease Investigator Group; Holmes JM, Manny RE, Lazar EL, Birch EE, Kelly KR, Summers AI, Martinson SR, Raghuram A, Colburn JD, Law C, Marsh JD, Bitner DP, Kraker RT, Wallace DK. A Randomized Trial of Binocular Dig Rush Game Treatment for Amblyopia in Children Aged 7 to 12 Years. Ophthalmology. 2019 Mar;126(3):456-466. doi: 10.1016/j.ophtha.2018.10.032. Epub 2018 Oct 22. PMID 30352226
- [Background] Birch EE, Morale SE, Jost RM, De La Cruz A, Kelly KR, Wang YZ, Bex PJ. Assessing Suppression in Amblyopic Children With a Dichoptic Eye Chart. Invest Ophthalmol Vis Sci. 2016 Oct 1;57(13):5649-5654. doi: 10.1167/iovs.16-19986. PMID 27784068
- [Background] Xiao S, Angjeli E, Wu HC, Gaier ED, Gomez S, Travers DA, Binenbaum G, Langer R, Hunter DG, Repka MX; Luminopia Pivotal Trial Group. Randomized Controlled Trial of a Dichoptic Digital Therapeutic for Amblyopia. Ophthalmology. 2022 Jan;129(1):77-85. doi: 10.1016/j.ophtha.2021.09.001. Epub 2021 Sep 14. PMID 34534556
- [Background] Martin S, Portela JA, Ding J, Ibarrondo O, Levi DM. Evaluation of a Virtual Reality implementation of a binocular imbalance test. PLoS One. 2020 Aug 21;15(8):e0238047. doi: 10.1371/journal.pone.0238047. eCollection 2020. PMID 32822405
- [Background] Li SL, Reynaud A, Hess RF, Wang YZ, Jost RM, Morale SE, De La Cruz A, Dao L, Stager D Jr, Birch EE. Dichoptic movie viewing treats childhood amblyopia. J AAPOS. 2015 Oct;19(5):401-5. doi: 10.1016/j.jaapos.2015.08.003. PMID 26486019
- [Background] Birch EE, Jost RM, De La Cruz A, Kelly KR, Beauchamp CL, Dao L, Stager D Jr, Leffler JN. Binocular amblyopia treatment with contrast-rebalanced movies. J AAPOS. 2019 Jun;23(3):160.e1-160.e5. doi: 10.1016/j.jaapos.2019.02.007. Epub 2019 May 16. PMID 31103562
- [Background] Manny RE, Holmes JM, Kraker RT, Li Z, Waters AL, Kelly KR, Kong L, Crouch ER, Lorenzana IJ, Alkharashi MS, Galvin JA, Rice ML, Melia BM, Cotter SA; Pediatric Eye Disease Investigator Group. A Randomized Trial of Binocular Dig Rush Game Treatment for Amblyopia in Children Aged 4 to 6 Years. Optom Vis Sci. 2022 Mar 1;99(3):213-227. doi: 10.1097/OPX.0000000000001867. PMID 35086119
- [Background] Sloper J. New Treatments for Amblyopia-To Patch or Play? JAMA Ophthalmol. 2016 Dec 1;134(12):1408-1410. doi: 10.1001/jamaophthalmol.2016.4296. No abstract available. PMID 27832261
- [Background] Liu XY, Zhang JY. Dichoptic training in adults with amblyopia: Additional stereoacuity gains over monocular training. Vision Res. 2018 Nov;152:84-90. doi: 10.1016/j.visres.2017.07.002. Epub 2017 Aug 4. PMID 28736224
- [Background] Liu XY, Zhang JY. Dichoptic De-Masking Learning in Adults With Amblyopia and Its Mechanisms. Invest Ophthalmol Vis Sci. 2019 Jul 1;60(8):2968-2977. doi: 10.1167/iovs.18-26483. PMID 31307059
- [Background] Liu XY, Zhang YW, Gao F, Chen F, Zhang JY. Dichoptic Perceptual Training in Children With Amblyopia With or Without Patching History. Invest Ophthalmol Vis Sci. 2021 May 3;62(6):4. doi: 10.1167/iovs.62.6.4. PMID 33944893
- [Background] Liu Z, Chen Z, Gao L, Liu M, Huang Y, Feng L, Yuan J, Deng D, Huang CB, Yu M. A New Dichoptic Training Strategy Leads to Better Cooperation Between the Two Eyes in Amblyopia. Front Neurosci. 2020 Nov 26;14:593119. doi: 10.3389/fnins.2020.593119. eCollection 2020. PMID 33324154
- [Background] Holmes JM, Manh VM, Lazar EL, Beck RW, Birch EE, Kraker RT, Crouch ER, Erzurum SA, Khuddus N, Summers AI, Wallace DK; Pediatric Eye Disease Investigator Group. Effect of a Binocular iPad Game vs Part-time Patching in Children Aged 5 to 12 Years With Amblyopia: A Randomized Clinical Trial. JAMA Ophthalmol. 2016 Dec 1;134(12):1391-1400. doi: 10.1001/jamaophthalmol.2016.4262. PMID 27812703
- See also: Visionary software webpage — http://www.visionarytool.com